CLINICAL TRIAL: NCT02427022
Title: Phase II Evidence-Based Practice in Community-Based Social Work: A Multi-Media Strategy
Brief Title: Implementation, Fidelity, and Outcomes Following Novel and Usual Critical Time Intervention Training
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Center for Social Innovation, Massachusetts (Other)
Collaborators: Columbia University (Other); Hunter College of City University of New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HHSN-271-2010-00032-C; HHSN-271-2010-00032-C (Other Grant/Funding Number: National Institute of Mental Health)
Record Dates: First submitted 2014-07-10; First posted 2015-04-27 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2014-07

CONDITIONS: Homeless Services; Human Services Training
Keywords: evidence based practices, critical time intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Online CTI Training (Experimental): Services providers in this group received a novel online CTI training. The enhanced course combines depth of knowledge among trainers, skills-based and practical approaches to learning, new technologies, and opportunities for social networking. The course is divided the knowledge, skills, and tools associated with CTI into four two-week modules. The total instruction time for the course was 24 hours.
  Interventions: Other: CTI
- Face-to-Face CTI Training (Active Comparator): Service providers in the group received 1.5-days of face-to-face CTI training at each study site with one trainer. There were a total of 8 hours of instructor led training per site. Face-to-face training sessions were followed by three assignments with feedback from trainers, and eight 60-minute telephone consultation sessions.
  Interventions: Other: CTI

INTERVENTIONS:
Other: CTI — CTI is an empirically supported, time-limited case management model designed to prevent homelessness and other adverse outcomes in people with mental illness following discharge from hospitals, shelters, prisons and other institutions. CTI was originally developed and tested by researchers and clinicians at Columbia University and New York State Psychiatric Institute with significant support from the National Institute of Mental Health and the New York State Office of Mental Health.

SUMMARY:
Clinical social workers and other staff providing direct care to individuals experiencing homelessness face multiple challenges in obtaining training and implementing evidence-based practices in diverse community settings. Critical Time Intervention (CTI) is an increasingly popular evidence based practice with these agencies.

With funding from a Phase II Small Business Innovation Research grant from the National Institute of Mental Health, the Center for Social Innovation developed an online multi-media training on CTI which incorporates a Community of Practice approach to encourage peer-based learning.

The primary aim of this longitudinal, randomized-control study is to compare and contrast this online training modality with a face-to-face training on implementation of and fidelity to the CTI model over time. Nearly two-hundred direct service providers from 20 homeless-service agencies were randomly assigned to complete either an online or face-to-face training in CTI. Pre-post training and knowledge-retention surveys, interviews with trainers, agency administrators, and providers were conducted to track satisfaction with the training and experiences in implementing CTI. CTI-specific chart forms are used to assess fidelity to the CTI model, and administrative data from the agencies capture client-level outcomes.

DETAILED DESCRIPTION:
In September 2008, the Center for Social Innovation (C4) was awarded a Small Business Innovation Research (SBIR) contract from the National Institute of Mental Health to test innovative ways to disseminate evidence-based practices (EBPs) in community settings. C4 selected the practice of Critical Time Intervention (CTI), a focused, time-limited case management model designed to prevent and end homelessness among people who have experienced mental illness, addiction, and trauma. CTI is widely recognized as an evidence-based practice. During Phase 1 of the project, C4 partnered with CTI experts at the Columbia University Mailman School of Public Health to develop and test a prototype version of an instructor-led online course that brought together live (synchronous) and multimedia self-paced (asynchronous) elements to train community-based social workers on the CTI model. The pilot study showed promising results in the areas of knowledge gain, knowledge retention, and confidence to implement the model. Based on these preliminary findings, C4 applied for Phase 2 funding, which was granted in September 2010.

Phase 2 of the study was completed in February 2013. This phase of the study included full product development of the online course and a randomized controlled trial comparing the online course with face-to-face CTI training (provided by our partners at the Center for Urban Community Services or CUCS). Specifically, the study included 179 service providers from 19 agencies across the United States and Canada. We randomly assigned each agency to one of two study conditions: 1) online training + community of practice, or 2) face-to-face training + telephone coaching. After they completed the training, we examined satisfaction with the training modalities, knowledge gains and knowledge retention. We then followed agencies' CTI implementation process and assessed CTI implementation readiness, experiences in implementing CTI, fidelity to the CTI model over time, and the impact of CTI implementation on the clients served by these agencies.

ELIGIBILITY:
Agency Inclusion Criteria:

1. Possessing administrative-level support for implementing CTI within the agency
2. Capability of engaging at least one CTI team in training
3. Willingness to engage in evaluation
4. A willingness to collect and share administrative client data

Agency Exclusion Criteria:

1. Not possessing administrative support
2. Not capable of of engaging at least one CTI team in training
3. Not willing to engage in evaluation
4. Not willing to collect and share administrative client data

Provider Inclusion Criteria:

1. Capacity to fill one of the three roles necessary for CTI team membership or eligibility to shift into those roles: Supervisor, Field Coordinator, or CTI Worker; and,
2. Willingness to engage in the CTI training and the study activities.

Provider Exclusion Criteria:

1. Individuals not working as a supervisor, field coordinator or CTI Worker within an eligible service organization.
2. Individuals not willing to engage in CTI training and study activities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2010-09; Primary Completion 2012-10 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change in confidence in CTI principles [attitudinal] | Pre and post surveys (June and July, 2011; weeks 1 and 2)
  Providers were asked to rate their confidence using a 5-point scale (1=not at all confident; 2=not really confident; 3=somewhat confident; 4=confident; 5=extremely confident) in eight key areas: 1) describing CTI as an intervention and its core principles; 2) describing who is on a CTI team and their roles; 3) describing the clinical treatment areas involved with CTI principles; 4) describing the five core skills of CTI and their purposes; 5) describing how to start a CTI program including identifying client and community needs; 6) identifying some of the challenges that might arise in trying to establish CTI in different settings; 7) how chart work differs from CTI work; and 8) describing the key indicators that CTi is implementing. Providers in both treatments were asked to complete these questions in both pre and post surveys.

SECONDARY OUTCOMES:
Training format preference [attitudinal] | Prior to intervention (June, 2011; week 1)
  After agencies were randomized and before training began, key informants within agencies were asked to participate in a semi-structure baseline interview where they were all asked what their preference was for training format.
Participant satisfaction [attitudinal] | Post interventions (July, 2011; week 2)
  Participant satisfaction was analyzed on the post survey and data were collected using a 3-point scale (1=not satisfied; 2=satisfied; 3=very satisfied).
Participant satisfaction [attitudinal] | Post intervention (March 2012; week 2)
  Participant satisfaction was also assessed qualitatively during follow-up interviews with a subset of providers.
Confidence in readiness to implement CTI principles [attitudinal] | Post intervention (June 2011; week 2)
  Providers were asked to rate their confidence in readiness to implement CTI principles in the post-survey and data were collected on a 5-point scale (1=not at all confident; 2=not very confident; 3=somewhat confident; 4=confident; and, 5= extremely confident) (see: Aarons, 2004).
Knowledge retention [knowledge] | Pre, post and follow up surveys weeks post training and six months post training (June 2011 and December 2011; weeks 1, 2 and 24)
  Providers who participated in both treatments were asked to complete a pre and post survey followed by a follow up survey in week 6 that looked for enduring effects attributable to participation in the study. Questions were posed in each of the key outcome areas listed above (1) describing CTI as an intervention and its core principles; 2) describing who is on a CTI team and their roles; 3) describing the clinical treatment areas involved with CTI principles; 4) describing the five core skills of CTI and their purposes; 5) describing how to start a CTI program including identifying client and community needs; 6) identifying some of the challenges that might arise in trying to establish CTI in different settings; 7) how chart work differs from CTI work; and 8) describing the key indicators that CTI is implementing).
Fidelity to CTI model | Post implementation (March 2012, June 2012, September 2012; weeks 40, 52, and 64)
  Providers completed modified version of CTI fidelity assessment paperwork based on that developed by CTI co-developer Sally Conover (see: da Silva, Lovisi & Conover, 2014). Using the CTI forms submitted by study sites, we assigned each provider a fidelity score. This score indicated how closely the providers' implementation of CTI aligned with the original model. Providers' fidelity scores were calculated based on:
  * Compliance Fidelity: The degree to which providers implemented the key CTI components, including: early engagement and early linking; working in the community; using a three-phased approach; focusing on only a few areas; completing the intervention within nine months.
  * Competence Fidelity: Measures how well intervention was documented, including quality and thoroughness of progress notes.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Olivet, MA, Principal Investigator — Center for Social Innovation
Locations (1):
- Center for Social Innovation, Needham, Massachusetts, United States

REFERENCES:
- [Background] da Silva, T. F. C., Lovisi, G. M. & Conover, S. (2014) Developing an instrument for assessing fidelity to the intervention in the Critical Time Intervention - Task Shifting (CTI-TS): Preliminary report. Archives of Psychiatry and Psychotherapy, 1: 55-62.
- [Background] Aarons GA. Mental health provider attitudes toward adoption of evidence-based practice: the Evidence-Based Practice Attitude Scale (EBPAS). Ment Health Serv Res. 2004 Jun;6(2):61-74. doi: 10.1023/b:mhsr.0000024351.12294.65. PMID 15224451